CLINICAL TRIAL: NCT00006185
Title: Cellular Mechanisms for Metabolic Dysfunction in HIV
Brief Title: Underlying Abnormalities in Fat and Muscle Leading to Lipodystrophy Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: hivtzd (completed); DK49316-06
Record Dates: First submitted 2000-08-22; First posted 2000-08-23 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections; Lipodystrophy; Insulin Resistance
Keywords: peripheral fat wasting; truncal adiposity; fat biopsy; muscle biopsy; intravenous lines; blood draws; insulin administration; sugar water; screening
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Insulin Resistance

INTERVENTIONS:
Drug: Avandia administration for 6-12 weeks

SUMMARY:
With the advent of highly active anti-retroviral therapy(HAART), patients with HIV disease are developing a series of metabolic abnormalities including peripheral fat wasting, increase in truncal fat, high serum triglyceride levels, insulin(a hormone that controls blood sugar) resistance with an increased incidence of Type 2 Diabetes Mellitus and elevated blood pressure. The premise of this study is that abnormalities in the ability of fat and muscle tissue to respond to the hormone insulin may be the cause of the diabetes mellitus, high serum triglyceride levels and abnormal fat distribution. The purpose of the study is to assess how insulin resistant patients with HIV disease are and if their fat and muscle tissue are responding abnormally to insulin. This is done by administering insulin and taking small tissue samples of fat and muscle from the upper thigh and assessing how good insulin acts in these tissues.

Patients with HIV disease will be admitted into the study after undergoing a screening medical history and examination. Once patients qualify, they will have their insulin resistance measured as well as the response of their fat and muscle to insulin; blood levels of glucose (sugar), cholesterol and triglycerides will be measured; body fat will be assessed using radiological tests; a detailed medical history will be obtained to assess risk factors for developing this syndrome.

Patients who are found to be insulin resistant will be offered a trial of an insulin sensitizing agent, called Avandia, for 6-12 weeks. It is hoped that the Avandia will restore the body's ability to respond normally to insulin (as it does in patients with Diabetes) and perhaps improve the fat abnormalities as well. All the same measures will be performed at the end of the course of Avandia as were done at baseline.

Patients who are not insulin resistant will be asked to come back yearly to assess whether they develop insulin resistance over time. This study will continue to recruit patients over the next 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosis of HIV or AIDS

Exclusion Criteria:

* Positive pregnancy test
* Diagnosis of cancer
* Acute illness (patients can be enrolled once stable)
* Hemoglobin less than 7.0 g/dl or acute heart problems
* Renal function greater than creatinine 1.5 mg/dl
* Liver dysfunction 3 times normal
* Use of medications like glucocorticoids and birth control pills
* Untreated hypertension
* Diabetes mellitus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Marie Gelato, Study Director — SUNY at Stony Brook
Locations (1):
- University Hospital at Stony Brook New York, Stony Brook, New York, United States